CLINICAL TRIAL: NCT02849860
Title: A Phase 1b Open-Label Study Evaluating the Absorption and Systematic Pharmacokinetics of Topically Applied IDP-121 Lotion in Subjects With Acne Vulgaris Under Maximal Use Conditions
Brief Title: Absorption and Systematic Pharmacokinetics of IDP-121 Lotion in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V01-121A-501
Record Dates: First submitted 2016-07-06; First posted 2016-07-29 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IDP-121 Lotion (Experimental): Lotion
  Interventions: Drug: IDP-121 Lotion

INTERVENTIONS:
Drug: IDP-121 Lotion — Lotion
  Other Names: Lotion

SUMMARY:
Open-Label study designed to assess the safety and plasma PK of tretinoin and relevant metabolites after topical dermal application of IDP-121 lotion.

DETAILED DESCRIPTION:
Open-Label study designed to assess the safety and plasma PK of tretinoin and relevant metabolites after topical dermal application of IDP-121 lotion in subjects with moderate to severe acne vulgaris under maximal use conditions.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, between the ages of 9 and <17 years (16 years 11 months inclusive).
* Written and oral informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or legal guardian must sign the informed consent.
* Subject must have a score of 3 (moderate) to 4 (severe) on the Evaluator's Global Severity Assessment at the screening and baseline visit in the facial area.
* Subjects with facial acne inflammatory lesions count no less than 20 but no more than 40.
* Subjects with facial acne non-inflammatory lesions count no less than 20 but no more than 100.

Key Exclusion Criteria:

* Use of investigational drug or device within 30 days of enrollment or participation in research study or concurrent study with this study.
* Any dermatological conditions on the face that could interfere with clinical evaluations acne conglobate, acne fulminans, secondary acne, perioral dermatitis, clinical significant rosacea, gram negative folliculitis.
* Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive.
* Subjects with facial beard or mustache that could interfere with any study assessments.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Evaluators Global Severity Score at Day 15 | 15 Days
  Acne severity will be determined by the investigator/evaluator based on a global assessment of the inflammatory and non-inflammatory lesions of facial acne. Evaluations will be graded on a static scale ranging from 0 (clear) to 4 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Valeant Pharmaceutical
Locations (2):
- United States (2):
  - Valeant Site 02, Austin, Texas
  - Valeant Site 01, College Station, Texas

IPD SHARING:
Plan to Share IPD: No